CLINICAL TRIAL: NCT00264940
Title: Diagnosis of Insulin Resistance: 13C-Glucose Breath Test Vs HOMA Index.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TASMC-05-ZH-315-CTIL
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2005-12-13 (Estimated); Status verified 2005-12

CONDITIONS: Glucose Intolerance; Insulin Resistance; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance; Diabetes Mellitus, Type 2

SUMMARY:
The prevalence of type 2 diabetes is rising in the population for many years. It is now recognized that a period of glucose intolerance precedes the clinical symptoms appearance. This is due to a combination of b-cell dysfunction and insulin resistance. It is estimated that this pre-clinical phase of type 2diabetes may antedate the onset of overt diabetes by 10-12 years. Furthermore, insulin resistance is considered to be a main component of the metabolic syndrome and associated with significant cardiovascular morbidity and mortality. Recently, there has been an effort to pinpoint the pre-diabetic phase for early therapeutic intervention in the individual. These studies, in patients with impaired glucose intolerance, have shown to be beneficial from both lifestyle change and pharmacological intervention. It is thus hypnotized that intervention in patients with insulin resistance with or without glucose intolerance may prevent the progress of type 2 diabetes and it's complications. There is difficulty in identifying individuals who are at high risk for type 2 diabetes. The prevention strategy relies on intervention in a pre-diseased state. In the case of type 2 diabetes, the early intervention is useful in the phase where there is insulin resistance, but prior to the appearance of glucose intolerance. The diagnosis of insulin resistance is a challenging one. The gold standard in diagnosing insulin resistance is the hyperinsulinemic-euglycemic clamp, but this method is not suitable for routine clinical use. Thus, less invasive methods for evaluation, like homeostasis model assessment (HOMA) and quantitative insulin sensitivity check index (QUICKI), were developed. There is a correlation between HOMA and QUICKI results and the hyperinsulinemic-euglycemic clamp. Both HOMA and QUICKI allow insulin resistance diagnosis. The results from those tests correlate with hyperinsulinemic-euglycemic clamp and allow diagnosing insulin resistance, however, those indexes require serum glucose, insulin measurements and quite complicated calculations. A new method was suggested, non-invasive, sensitive and simple, for the identification of insulin resistance. In normal individuals, in the presence of insulin, glucose is taken up by a variety of cells, undergoes glycolysis and enters the tricarboxylic acid cycle or fat synthesis. In either case, CO2 in produced as a by-product. This CO2 enters the circulation and is discarded by the lungs. The new method is based on the assumption that 13C-glucose is ingested as described and its by-product 13CO2 can be measured in the expired air. In type 2 diabetes and other states of insulin resistance glucose, uptake is impaired and results in blunted 13CO2 production. This hypothesis was tested by Lewanczuc et al. The writers compared the [13C]-glucose breath test with hyperinsulinemic-euglycemic clamp, HOMA and QUICKI indexes. They tested 26 patients at different stages of insulin sensitivity and reported a good correlation of the glucose breath test and the other indexes. We suggest testing a larger group of patients at high-risk to develop type 2 diabetes and compare the glucose breath test with HOMA index.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to fast over night
* A blood sample should be drawn

Exclusion Criteria:

* Insulin dependent diabetes
* Pulmunary disorder
* Gastrointestinal disorder
* Endocrine disorder

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Zamir Halprn, MD, Study Chair; Ilana Goldiner, PhD, Principal Investigator; Yochanan Peled, PhD, Principal Investigator